CLINICAL TRIAL: NCT02596919
Title: Fast Infrared Meibography (Photography)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After review, recruitment was halted as the images obtained needed improvement. To be presented at the British Oculoplastic Surgery Society in Jun 17
Sponsor: Queen Victoria Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RPC302
Record Dates: First submitted 2015-08-13; First posted 2015-11-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Photography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No arms (Other): No randomisation therefore no arms. All patients will receive the same research treatment.
  Interventions: Other: photography

INTERVENTIONS:
Other: photography — photography of meibomian glands

SUMMARY:
Infrared meibography is a useful technique in the evaluation of meibomian gland disease (MGD). MGD is a major cause of dry eye symptoms, affecting a large number of patients seen in the Corneo-Plastic Unit (CPU). Many parameters have been used to evaluate MGD including tear film break-up time, lid margin abnormalities, and Schirmer tear test values. Direct visualization of meibomian glands by infrared meibography has been shown to correlate well with these parameters.

Although infrared meibography was developed more than 30 years ago, it is not widely used. This has probably been due to the need for special equipment, examiner time and expertise and patient discomfort during the examination. Analysis of the acquired images also needed to be from video review with extraction of video stills - a time-consuming process.

Investigators aim to pilot a rapid non-contact (non-painful) method of obtaining infrared images of meibomian glands using equipment already available at QVH. This pilot study will validate the technique and check patient acceptability. Investigators are hopeful this test could be used as a useful tool for future research into dry eye conditions and MGD.

DETAILED DESCRIPTION:
Patients will receive a patient information sheet in the post with their Eye Clinic appointment letter. To be clear, the points listed below would form the standard of care for a dry eye patient attending the clinic, apart from the additional infrared photographic image taken for the study (point 6).

In the Consultation room, the study will be explained to participants by one of the investigators. If they agree to participate, a consent form will be signed by the participant and an investigator. They will be questioned regarding the absence or presence of ocular symptoms using a previously validated and accepted scoring scale (Ocular Surface Disease Index - OSDI). This questionnaire will allow patients to score their degree of dry eye symptoms.

Participants will then undergo:

1. Schirmers tear test of production.
2. Clinical slit lamp examination to look for abnormalities of the upper and lower lid margins.
3. Fluorescein staining of the ocular surface (divided into 3 zones comprising nasal conjunctival, corneal, and temporal conjunctival areas).
4. Observation of tear film break-up time (TBUT).
5. Digital pressure was applied to the upper tarsus, and the degree of ease with which meibomian secretion (meibum) is induced, evaluated semi-quantitatively. Eversion of upper and lower eyelids in the clinic is part of the standard ocular examination.
6. In the photography department, the upper and lower eyelids will then be everted and non-contact infrared photographs taken. Partial or complete loss of Meibomian glands will be scored according to the meiboscore for each eyelid. After the image is taken, patient experience will be gathered on a five-point Lickert scale score sheet.

Outcome measures To examine for a correlation between morphologic changes in meibomian glands visible on infrared photography and both clinical examination findings and questionnaire scores regarding eyelid and tear film function in the population.

To assess patient experience and acceptability of the intervention.

4.0 Selection and withdrawal of Subjects 4.1 Inclusion criteria

Patients attending the CPU will be offered the opportunity to take part if they comply with the following:

* Over 18 years of age
* Able to give their informed consent

4.2 Exclusion criteria:

* Patients under the age of 18 years of age
* Poor understanding of language
* Ocular allergies
* History of contact lens wear
* History of eye or eyelid surgery
* Systemic or ocular diseases that may interfere with tear film production or function.
* Use of systemic medication with tetracycline derivatives, antihistamines, isotretinoin, or nutritional supplements for MGD.
* Use of topical ciclosporin-A or steroids beginning within the last month.
* Refusal for patient's own GP to be informed of participation.

5.0 Treatment of subjects Participants will undergo the standard of care in the Corneo-Plastic Unit, but will also be examined and photographed by the infrared technique.

6.0 Assessment of Efficacy Through the assessment described above, a statistical analysis between OSDI score, ocular surface and Meibomian gland score will be possible. We will analyse the findings to see if there is any relationship between the patient symptoms and level of Meibomian gland dysfunction.

7.0 Assessment of Safety Any side effects reported by the patient and/or observed by the clinician will be recorded. Data regarding patient experience of the test will also be collected.

ELIGIBILITY:
Inclusion criteria

Patients attending the CPU will be offered the opportunity to take part if they comply with the following:

* Over 18 years of age
* Able to give their informed consent

Exclusion criteria:

* Patients under the age of 18 years of age
* Poor understanding of language
* Ocular allergies
* History of contact lens wear
* History of eye or eyelid surgery
* Systemic or ocular diseases that may interfere with tear film production or function.
* Use of systemic medication with tetracycline derivatives, antihistamines, isotretinoin, or nutritional supplements for MGD.
* Use of topical ciclosporin-A or steroids beginning within the last month.
* Refusal for patient's own GP to be informed of participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To examine for a correlation between morphologic changes in meibomian glands visible on infrared photography with clinical examination findings | 5 minutes
  To examine for a correlation between morphologic changes in meibomian glands visible on infrared photography and both clinical examination findings and questionnaire scores regarding eyelid and tear film function in the population. Schirmer 1 Tear Test A Schirmer 1 test evaluates baseline secretion.
  1. 0.5% proxymetacaine eye drops are administered to achieve topical anaesthesia.
  2. Schirmer strips are then inserted into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding corneal touch.
  3. All patients are seated at rest with their eyes closed.
  4. The length of wetting strips in millimeters is recorded after 5 minutes.
  The Schirmer Test is interpreted after 5 minutes as follows:
  * Normal aqueous tear production is supported by measurements of > 15 mm.
  * Mild-moderate reduction of aqueous production: 5mm-14mm.
  * Severe dryness due to reduced tear production is < 5mm.

SECONDARY OUTCOMES:
To examine for a correlation between morphologic changes in meibomian glands visible on infrared photography with questionnaire scores | 5 minutes
  OSDI Questionnaire (OSDI) - A validated and accepted scoring scale, with scores ranging from 0 (None of the time) to 4 (All of the time).

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Victoria Hospital NHS Foundation Trust, East Grinstead, W Sussex, United Kingdom